CLINICAL TRIAL: NCT05266885
Title: Prevalence of Hypertension in Type-2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Kabul University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Habib Ahmad Esmat, Research committee, Kabul University of Medical Sciences
Other Study IDs: 0003
Record Dates: First submitted 2022-02-20; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Prevalence of Elevated Blood Pressure in Type-2 Diabetics
Keywords: Prevalence; Hypertension; Type-2 diabetes
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male and Female: (37 male, 63 female)

SUMMARY:
Cardiovascular disease is the most prevalent cause of morbidity and mortality in diabetic patients. Hypertension has been confirmed as a major risk factor for cardiovascular disease, which is frequently associated with diabetes mellitus. Therefore, the detection and management of elevated blood pressure (BP) is a critical component of the comprehensive clinical management of diabetics. Since the rates of hypertension in diabetics are lacking in Afghanistan, this study aimed to evaluate the prevalence of elevated blood pressure in type-2 diabetic patients.

DETAILED DESCRIPTION:
Cardiovascular disease is the most prevalent cause of morbidity and mortality in diabetic patients. Hypertension has been confirmed as a major risk factor for cardiovascular disease, which is frequently associated with diabetes mellitus. Therefore, the detection and management of elevated blood pressure (BP) is a critical component of the comprehensive clinical management of diabetics. Since the rates of hypertension in diabetics are lacking in Afghanistan, this study aimed to evaluate the prevalence of elevated blood pressure in type-2 diabetic patients.

This is a descriptive cross-sectional study, which included 322 type -2 diabetic patients (37 male, 63 female) who were presented to our center from November 2019 to January 2020.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed diabetic patients
* Newly diagnosed Diabetics
* known case of diabetes

Exclusion Criteria:

* The patients who were seriously ill
* Pregnant women
* Type-1 diabetic patients,

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Type -2 diabetics who were presented to our center from November 2019 to January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
High incidence of HTN in Diabetics | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad wali Nasary, MD, Principal Investigator — KMUs
Locations (1):
- Habib Ahmad Esmat, Kabul, None Selected, Afghanistan

IPD SHARING:
Plan to Share IPD: Undecided